CLINICAL TRIAL: NCT01678430
Title: A Randomised Investigation of Alternative Ofatumumab-containing Regimens in Less Fit Patients With CLL
Brief Title: A Trial Looking at Ofatumumab for People With Chronic Lymphocytic Leukaemia Who Cannot Have More Intensive Treatment
Acronym: RIAltO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Liverpool (Other)
Collaborators: GlaxoSmithKline (Industry); Napp Pharmaceuticals Limited (Industry); Chugai Pharma USA (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OMB114578; 2011-000919-22 (EudraCT Number); 009988575 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2012-08-30; First posted 2012-09-05 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-08

CONDITIONS: Chronic Lymphocytic Leukaemia
Keywords: Chronic Lymphocytic Leukaemia; Less fit; CD20 antibody; Ofatumumab; Chlorambucil; Bendamustine
MeSH Terms: conditions — Leukemia, B-Cell | interventions — ofatumumab; Chlorambucil; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ofatumumab-Chlorambucil (Active Comparator): Ofatumumab cycle 1: 300mg iv day 1, 1000mg iv day 8; cycle 2 onwards: 1000mg iv day 1 Chlorambucil: 10mg/m2 po days 1-7
  Interventions: Drug: Ofatumumab; Drug: Chlorambucil
- Ofatumumab-Bendamustine (Experimental): Ofatumumab cycle 1: 300mg iv day 1, 1000mg iv day 8; cycle 2 onwards: 1000mg iv day 1 Bendamustine: 70mg/m2 iv days 1 and 2
  Interventions: Drug: Ofatumumab; Drug: Bendamustine

INTERVENTIONS:
Drug: Ofatumumab
  Other Names: Arzerra
Drug: Chlorambucil
  Other Names: Leukeran
  Arms: Ofatumumab-Chlorambucil
Drug: Bendamustine
  Other Names: Levact
  Arms: Ofatumumab-Bendamustine

SUMMARY:
The purpose of this study is to compare ofatumumab & chlorambucil (O-Chl) versus ofatumumab & bendamustine (O-B) in patients with Chronic Lymphocytic Leukaemia who are considered not fit enough for rituximab, fludarabine & cyclophosphamide (R-FC).

DETAILED DESCRIPTION:
Chlorambucil (Chl) has been the mainstay of CLL treatment for half a century. However, frontline treatment has improved considerably over the last decade, first by the advent of fludarabine plus cyclophosphamide (FC), and more recently by the addition of the anti-CD20 antibody, rituximab, to FC. Although FC-based regimens are considerably more effective than Chl, they are also associated with greater toxicity which makes them inappropriate for less fit patients. This is an important consideration, given that CLL predominantly affects older people who tend to have more co-morbidity. Although a single-arm phase II study (Roche MO20927; NCRI CLL208) has shown that R-Chl is safe and effective, there are no phase III data proving the benefit of adding an anti-CD20 antibody to Chl. This question is currently being addressed by a phase III RCT of Chl with or without ofatumumab (GSK OMB110911 / COMPLEMENT-1 / NCRI CLL7). Ofatumumab is a fully human anti-CD20 antibody that binds to an epitope distinct from that of rituximab and produces more complement-dependent cytotoxicity. The RIAltO trial is a direct follow-on to the NCRI CLL7 phase III RCT trial in less fit patients and therefore the Ofatumumab dose has been selected to mirror the regimen used in that trial.

ELIGIBILITY:
Inclusion Criteria:

1. CLL/SLL requiring treatment by NCI/IWCLL 2008 criteria. At least one of the following criteria:

   1. Progressive marrow failure as manifested by the development of, or worsening of, anaemia and/or thrombocytopenia.
   2. Massive (i.e. 6 cm below the left costal margin) or progressive or symptomatic splenomegaly.
   3. Massive (i.e. 10 cm in longest diameter) or progressive or symptomatic lymphadenopathy.
   4. Progressive lymphocytosis with an increase of more than 50% over a 2-month period or lymphocyte doubling time (LDT) of less than 6 months.
2. No prior cytotoxic or targeted therapy for CLL
3. Full-dose R-FC considered inappropriate for at least one of the following reasons

   1. Age 75 or greater
   2. WHO performance status 2 or 3
   3. Cardiac impairment (NYHA class II)
   4. Respiratory impairment (bronchiectasis or moderate COPD)
   5. Renal impairment (estimated Glomerular Filtration Rate (eGFR) 10-30 ml/min)
   6. Any other significant co-morbidity or factor that makes R-FC inappropriate
4. Considered able to tolerate Chl at the dose used in the LRF CLL4 trial (10mg/m2 d1-7)
5. Written informed consent

Exclusion Criteria:

1. Neutrophil count less than 1.0 x 109/l or platelet count less than 50 x 109/l unless due to CLL
2. Uncontrolled auto-immune haemolytic anaemia or thrombocytopenia
3. Active infection
4. Seropositivity for HIV, HCV or HBV (surface antigen or and core antibody)
5. Severe renal impairment (eGFR less than 10ml/min)
6. Severe hepatic impairment (serum bilirubin more than twice the upper limit of normal) unless due to CLL or Gilbert's syndrome.
7. Concurrent treatment with glucocorticoids equivalent to more than prednisolone 20mg od
8. Prior treatment with monoclonal antibody therapy within the last 3 months.
9. Yellow fever vaccination within 4 weeks prior to treatment start
10. Known hypersensitivity to ofatumumab, bendamustine or chlorambucil or any of their excipients
11. CNS involvement with CLL
12. History of Richter transformation
13. Concomitant malignancies within the last 3 years except successfully treated non-melanoma skin cancer or carcinoma in situ.
14. Major surgery within 28 days prior to randomisation
15. WHO performance status 4
16. Severe cardiac disease including unstable angina, acute myocardial infarction within six months prior to randomization, congestive heart failure (NYHA III-IV), and arrhythmia (excluding extra systoles or minor conduction abnormalities) unless controlled by therapy.
17. Any serious underlying medical or psychological conditions, which could impair the ability of the patient to participate in the trial or compromise ability to give informed consent
18. Treatment within a clinical trial within 30 days prior to trial entry.
19. Adult patient under tutelage (not competent to sign informed consent).
20. Pregnant or lactating women.
21. Women of childbearing potential, including women whose last menstrual period was less than one year prior to screening, unable or unwilling to use adequate contraception from study start to one year after the last dose of protocol therapy. Adequate contraception is defined as hormonal birth control, intrauterine device, double barrier method or total abstinence.
22. Male subjects unable or unwilling to use adequate contraception methods from study start to one year after the last dose of protocol therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 670 (Estimated)
Dates: Start 2011-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | There are three pre-planned analyses of the PFS primary endpoint: end recruitment (approx 150 events); 300 events (after a minimum 12 months follow up for all patients), 400 events (after a minimum 24 months follow up for all patients)
  Calculated from the date of randomisation to the date of progression or death, or the censor date.

SECONDARY OUTCOMES:
Duration of response | 6 years (after 2 years follow up of the last patient recruited)
  Response duration is defined as the time from when the criteria for partial or complete response are met until the first documentation of relapse or progression.
Overall survival | 6 years (after 2 year follow up of the last patient recruited)
  Overall survival is defined as the time from initiation of study treatment to death, irrespective of cause or subsequent treatment. Patients still alive at the time of analysis will be censored at the date last seen alive at last follow up.
Time to treatment failure | 6 years (after 2 year follow up of the last patient recruited)
  Time to treatment failure is defined as the time from initiation of study treatment to death, disease progression, or initiation of alternative treatment due to failure to achieve a complete or partial response to the study treatment.
Toxicity | 6 years (after 2 years follow up of the last patient recruited)
  Haematological toxicity will be reported in accordance with the 2008 NCI/IWCLL guidelines. Non-haematological toxicity will be reported in accordance with the current Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.
Treatment dose administered | 5 years (assuming last patient in receives 12 cycles of treatment)
  The number of cycles of treatment and cumulative dose of individual drugs administered will be summarised for each treatment group separately and compared across treatment groups
Quality of life | 6 years (after 2 years follow up of the last patient recruited)
  Quality of life will be assessed using the EQ-5D; EQ-VAS; EORTC QLQ-C30 and EORTC QLQ-CLL16 questionnaires. To standardise the raw scores, they will be linearly transformed into 0-to-100 scores.
Health Economic analysis | 6 years (after 2 years follow up of the last patient recruited)
  The economic evaluation will take the form of a cost-effectiveness analysis with the differential cost of the alternative treatments will be related to their differential benefits in terms of quality-adjusted life years (QALYs). Incremental cost-utility ratios will be estimated based on QALY estimates.
  A range of uni- and multi-variate, as well as probabilistic sensitivity analyses will be conducted to assess the robustness of the analysis.
  The use of bootstrapping and cost-effectiveness acceptability curves will facilitate a measure of variability around cost-effectiveness estimates. Sensitivity analysis will be used to consider the importance of sources of uncertainty other than sample variation (e.g. unit costs, discount rates).
  A model-based extrapolation of the trial results will be performed to explore the impact of a longer analytic time horizon, and consideration of health outcomes on the treatment cost-effectiveness.
Analysis of frailty and co-morbidity | Baseline, 2 months post treatment
  Patients outcomes will be compared across patient subgroups defined by CIRS, performance status, Vulnerable Elders Survey-13, Groningen Frailty Index (GFI) questionnaires and the Timed 'Up and Go' test.
Predictive value of biomarkers | Baseline, every 6 months until 42 months from study entry, disease progression
  Patient outcomes will be compared across patient subgroups defined by clinical (e.g. age, sex, stage) and laboratory (e.g. chromosomal, abnormalities, IGHV mutation status, TP53 mutation status).
Response | Baseline; 2 months post treatment; 6 months post treatment
  Response following initial therapy will be assessed in accordance with the revised (2008) NCI/IWCLL response criteria applicable to CLL. Minimal residual disease will be assessed by multicolour flow cytometric analysis of bone marrow aspirate samples taken 2 months after completing treatment and of blood samples taken 2 and 6 months after completing treatment.

CONTACTS AND LOCATIONS:
Locations (28):
- United Kingdom (28):
  - Countess of Chester Hospital, Chester, Cheshire
  - Derriford Hospital, Plymouth, Devon
  - Torbay Hospital, Torquay, Devon
  - Royal Bournemouth Hospital, Bournemouth, Dorset
  - Dorset County Hospital, Dorchester, Dorset
  - Colchester General Hospital, Colchester, Essex
  - Basingstoke and North Hampshire Hospital, Basingstoke, Hampshire
  - Southampton General Hospital, Southampton, Hampshire
  - Barnet and Chase Farm Hospitals, Enfield, Hertfordshire
  - Kent and Canterbury Hospital, Canterbury, Kent
  - Maidstone Hospital, Maidstone, Kent
  - Princess Royal Hospital, Orpington, Kent
  - Queen Elizabeth Hospital, Woolwich, London
  - West Middlesex University Hospital, Isleworth, Middlesex
  - Ealing Hospital, Southall, Middlesex
  - Hillingdon Hospital, Uxbridge, Middlesex
  - Belfast City Hospital, Belfast, Northern Ireland
  - Royal United Hospital, Bath, Somerset
  - Weston General Hospital, Weston-super-Mare, Somerset
  - Queens Hospital, Burton-on-Trent, Staffordshire
  - Queen Elizabeth Hospital, Gateshead, Tyne and Wear
  - Queen Elizabeth Hospital, Birmingham, West Midlands
  - Bradford Royal Infirmary, Bradford, West Yorkshire
  - Airdale General Hospital, Keighley, West Yorkshire
  - St James University Hospital, Leeds, West Yorkshire
  - Salisbury District Hospital, Salisbury, Wiltshire
  - Arrowe Park Hospital, Upton, Wirral
  - Royal Liverpool Hospital, Liverpool

REFERENCES:
- [Derived] Lim YJ, Duckworth AD, Clarke K, Kennedy P, Karpha I, Oates M, Gornall M, Kalakonda N, Slupsky JR, Pettitt AR. Influence of polyfunctional Tbet+ T cells on specific clinical events in chronic lymphocytic leukaemia. Front Immunol. 2025 Apr 17;16:1528405. doi: 10.3389/fimmu.2025.1528405. eCollection 2025. PMID 40313965
- See also: ISRCTN — http://www.controlled-trials.com/ISRCTN09988575/bendamustine
- See also: CancerHelp UK — http://cancerhelp.cancerresearchuk.org/trials/trials-search/a-trial-looking-ofatumumab-people-chronic-lymphocytic-leukaemia-who-cannot-have-more-intensive-treatment-rialto